CLINICAL TRIAL: NCT02172859
Title: Dietary Influence on Serotonin in Cognitive and Emotional Functioning in Women Using a Tryptophan-rich Protein Over 19 Days
Brief Title: Dietary Influence on Serotonin in Cognitive and Emotional Functioning in Women
Acronym: P2B_UK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: P2B-05
Record Dates: First submitted 2014-06-23; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
Keywords: lumiVida™, cognition, mood, sleep, tryptophane
MeSH Terms: interventions — LumiVida

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- lumiVida™ (Active Comparator): lumiVida™ (2 x 0.5 g sachets to be dissolved in 150ml water/ day): First dose 2h after breakfast and second dose 60-90min before bed-time for 19 days.
  Interventions: Dietary Supplement: lumiVida™
- Placebo (Placebo Comparator): Placebo (2 x 0.5 g sachets of casein hydrolysate to be dissolved in 150ml water/ day): First dose 2h after breakfast and second dose 60-90min before bed-time for 19 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: lumiVida™
  Arms: lumiVida™
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether a chronic dose of a tryptophan-rich protein drink (lumiVida™) can improve cognitive function, emotional processing and sleep in middle-aged women. In addition, also genetic predictors of susceptibility to an increase of Trp levels will be investigated.

lumiVida™ is considered a dietary supplement, and therefore it is not an approved drug by the Food and Drug Administration (FDA). It is regulated like a food. The U.S. Food and Drug Administration does not strictly regulate herbs and dietary supplements. The investigators do not claim that this supplement is meant to treat any ailment

DETAILED DESCRIPTION:
The treatment conditions are either placebo or lumiVida™ (N=30 per group) 0.5 g twice a day (total 1 g/ day). The first testing took place on the screening day (baseline). Subsequently, participants were supplied with supplements for 19 days intervention (sachets which had to be dissolved in 200-ml water). After 19 days, participants were tested again (same tests as on the baseline day). An additional facet was the completion of a 'sleep diary', which asks questions about sleep quality and latency, and bed-time mood, as well as allowing recording of timing of supplement taking.

ELIGIBILITY:
Inclusion Criteria:

* Physically and mentally healthy (defined by not concurrently receiving medical/pharmacological treatment (except mild painkillers), free of gastrointestinal complaints, not in pain, not diagnosed with a psychiatric disorder
* Female
* Aged: 45 - 65 years

Exclusion Criteria:

* Having received treatment in the last 12 months for: depression, anxiety, neurological disease including migraine, dementia, epilepsy, Parkinson's.
* History of any psychiatric or neurological illness in the last 2 years.
* Current medication targeting the brain (except mild painkillers, e.g. pure paracetamol, ibuprofen), including steroids, e.g. for contraception, Hormone Replacement Therapy (HRT), drugs for weight control, stimulants (e.g. phenylephrine, ephedrine), antihistamines, and some herbal or nutritional remedies including St. John's Wort, 5-hydroxy-tryptophan, or melatonin (which can affect the serotonin system).
* Pregnancy
* Current gastrointestinal complaints
* Diabetes (Type 1 or 2)
* Body mass index < 18 or > 35

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2010-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in measures of mood (MAPS scale) at day 19 | Day1 (baseline) and day 19
  Computer-based series of 9-point ratings scales to measure mood
Change from baseline in sleep diaries until day 19 | Day 1 and 2 prior treatment (baseline) and at day 1, 2, 4, 5, 11, 12, 18 and 19 of intake period
  Sleep diaries: Questions about sleep quality and latency, bed-time mood and alertness aspects.
Change from baseline in "Simple Reaction Time (SRT)" at day 19 | Day 1 (baseline) and day 19
  Measurement of reaction time and sustained attention
Change from baseline in the "Rotary Pursuit Task" at day 19 | Day 1 (baseline) and day 19
  Measurement of psychomotor coordination and motor learning
Change from baseline in "Verbal Recognition Memory test (VRM)" at day 19 | Day 1 (baseline) and day 19
  Recognition of words out of a list of words they have seen before
Change from baseline in "Match To Sample Visual search (MTS)" at day 19 | Day 1 (baseline) and day 19
  Measurement of visual attention, and speed and accuracy of responding
Change from baseline in "Rapid Visual Information Processing task (RVIP)" at day 19 | Day 1 (baseline) and at day 19
  Assessment of sustained attention and working memory
Change from baseline in "Affective Go/No-Go" at day 19 | Day 1 (baseline) and day 19
  Assessment of information processing biases for positive and negative stimuli
Change from baseline in "Emotion Recognition Task" at day 19 | Day 1 (baseline) and day 19
  Assessment of relatively enhanced recognition of positive emotional facial expressions on "morphed" photographs
Change from baseline in "Driving Hazard Perception Test" at day 19 | Day 1 (baseline) and day 19
  Measurement of participant's ability to perceive accurately and react to potential hazards whilst driving: this will be measured by computer software that displays a video recording from the driver's perspective through the windscreen of a moving car.

SECONDARY OUTCOMES:
Genetic evaluation of genotypes of the serotonin transporter protein (5HTTP) | Baseline
  Buccal (cheek) cell assays for DNA extraction for 5HTTP polymorphism analysis
Change from baseline in plasma TRP/LNAA ratio at day 19 | Day 1 (baseline) and day 19
  Measurement of L-tryptophan (TRP) and large neutral amino acids (LNAA) amino acids in blood samples (plasma)

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Gibson, Dr., Principal Investigator — School of Human & Life Sciences, Roehampton University, Holybourne Avenue London SW15 4JD, UK
Locations (1):
- School of Human & Life Sciences, London, London, United Kingdom

REFERENCES:
- [Background] Leigh Gibson E, Green MW. Nutritional influences on cognitive function: mechanisms of susceptibility. Nutr Res Rev. 2002 Jun;15(1):169-206. doi: 10.1079/NRR200131. PMID 19087403